CLINICAL TRIAL: NCT06916052
Title: An Observational Study of the Digital Platform Use for the Preparation and Monitoring of Patients With Scheduled Outpatient Colonoscopy
Brief Title: Study to Analyse the Use of a Digital Platform for the Preparation and Follow-up of Patients With Scheduled Outpatients Colonoscopy
Acronym: COLObs
Status: Recruiting | Type: Observational
Sponsor: Persei Vivarium (Other)
Collaborators: Effice Servicios Para la Investigacion S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: COLObs
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Outpatient Colonoscopy
Keywords: Colonoscopy preparation; Digital Platform; Caaring; Outpatient colonoscopy; DTx; Patient-reported Data; Real World Data; RWD; PROMs; Digital Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this clinical trial investigation with device is to to analyze the use of the Caaring® digital platform for the preparation and follow-up of scheduled colonoscopy.

Colonoscopy is a difficult procedure, and it is estimated that bowel preparation is inadequate in about 25% of patients. The main question it aims to answer is if the use of a digital platform (Caaring®) could be an effective tool for reducing the percentage of inadequate bowel preparations in patients with a scheduled colonoscopy. To this end, the application will provide precise instructions to patients.

A prospective, single-center, observational study with software device: The recruitment phase is expected to last two months. Patients will be followed for one month after the colonoscopy and 14 days prior to it.

Additionally, measuring patient experience and monitoring adverse effects after a colonoscopy are crucial to improving the safety of colonoscopies and the quality of healthcare, promoting higher quality colonoscopy services.

For that to happen, participants must have sufficient technological skills to use a smartphone.

DETAILED DESCRIPTION:
A prospective, single-center, observational study with software device. The protocol and informed consent documents have been reviewed and approved by the hospital human subjects reviewboard and the study will be performed in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Signed informed consent.
* Patients scheduled for outpatient colonoscopy.
* Patients able to complete the study questionnaires.
* Patients who regularly use a smartphone

Exclusion Criteria:

* Patients enrolled in the population-based colorectal cancer screening program with a positive fecal occult blood test.
* Minors or elderly patients (over 80 years of age).
* Patients with prior colorectal surgery.
* Patients who, in the opinion of the researcher, will not be able to commit to follow-up or lack adequate technological skills.
* Inability to provide adequate informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the Hospital Clínic in Barcelona diagnosed with a scheduled colonoscopy who meet the selection criteria and sign the informed consent will be included.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients scheduled colonoscopy who have an adequate bowel preparation. | Day 0, (Colonoscopy Day)
  Percentage of colonoscopies with adequate bowel preparation defined as having a total Boston Bowel Preparation Scale (BBPS) score greater than or equal of 6 and BBPS score for per colon segment ≥2.

SECONDARY OUTCOMES:
Active Patient Rate | Day -14 (14 days before the colonoscopy)
  Active patient rate defined as the number of patients who activate their account divided by the total number of patients guests.
Patients with section completed: Treatments | Day -14 (14 days before the colonoscopy)
  Of active patients, percentage who completes the section Treatments
Patients with section completed: Pick up the bowel preparation | Day -10 (10 days before colonoscopy)
  Of active patients, percentage who completes the section Pick up the bowel preparation.
Patients with section completed: Colonoscopy Preparation Solution (laxative). | Day 2 (2 days after colonoscopy)
  Of active patients, percentage who completes the secion Colonoscopy Preparation Solution (laxative).
Patients with section completed: Procedure satisfaction questionnaire | Day 3 (3 days after colonoscopy)
  Of active patients, percentage who completed the section Procedure satisfaction questionnaire.
Patients with section completed: Adverse Events | Day 1, Day 14 and Day 30
  Of active patients, percentage of patients who completes the Adverse Events section.
Percentage of patients with 100% of data completed | Day 31 (31days after the colonoscopy)
  Percentage of patients with 100% of data completed in the application.
Patients who view educational materials: Pick up the laxative | Day -10 (10 days before colonoscopy)
  Of active patients, percentage of Patients who view the educational materials: Pick up the laxative. The app will reflect the date and time that patients viewed that information.
Patients who view educational materials: Diet | Day -4 (4 days before colonoscopy)
  Of active patients, percentage of Patients who view the educational material: Diet. The app will reflect the date and time that patients viewed that information.
Patients who view educational materials: Adequate preparation for a colonoscopy | Day -4 (4 days before colonoscopy)
  Of active patients, percentage of Patients who view the educational material: Adequate preparation for a colonoscopy . The app will reflect the date and time that patients viewed that information.
Patients who view educational materials: Bring someone | Day -4 (4 days before colonoscopy)
  Of active patients, percentage of Patients who view the educational material: bring someone. The app will reflect the date and time that patients viewed that information.
Patients who view educational materials: Instructions for your colonoscopy | Day -3 (3 days before colonoscopy)
  Of active patients, percentage of Patients who view the educational material: Instructions for your colonoscopy. The app will reflect the date and time that patients viewed that information.
Percentage of patients with 100% of education materials viewed. | Day 31 (31days after the colonoscopy)
  Percentage of patients with 100% of educational materials viewed in the application.
Percentage of patients who take the laxative | Day -3 (3 days before the colonoscopy)
  Percentage of patients who take the laxative.
Patient satisfaction with the bowel preparation (laxative) | Day 2 (2 days after colonoscopy)
  The patient satisfaction with the bowel preparation will be measured through a specific satisfaction questionnaire created for this purpose. (Value 1-4). A higher score reflects greater satisfaction with software care.
Patient satisfaction with the colonoscopy experience | Day 3 (3 days after colonoscopy)
  The patient satisfaction with the colonoscopy experience will be measured through a specific satisfaction questionnaire created for this purpose. (Value 1-5). A higher score reflects greater satisfaction with software care.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No